CLINICAL TRIAL: NCT03894748
Title: A Parallel, Randomized, Double Blind, Multi-center, Active Drug Controlled, Phase III Clinical Trial to Compare the Efficacy and Safety of MT10109L Versus BOTOX® in Treatment of Glabella Line(Including a Preliminary Study to Evaluate Safety of MT10109L)
Brief Title: Efficacy and Safety Study of MT10109L in the Treatment of Glabella Line(Including a Preliminary Study to Evaluate Safety of MT10109L)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT_PRT_GL02
Record Dates: First submitted 2012-04-24; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Glabella Line Severity
Keywords: Glabella line; Glabella lines; Botulinum Toxin
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MT10109L(Botulinum toxin type A) (Experimental)
  Interventions: Drug: Botulinum Toxin Type A
- BOTOX® 50U(Botulinum toxin type A) (Active Comparator)
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — 20U of the investigational drug will be intramuscularly injected to 5 sites of the glabella line. Treatment will be conducted just once in visit 2.

SUMMARY:
This study design is multi-center, randomized, double-blind, parallel group, active controlled, phase 3 clinical trial(Including randomized, double-blind, parallel group, active controlled, preliminary study). Subjects who voluntarily signed the informed consent and are judged to be eligible for this study will be intramuscularly injected with the study drug or the comparator at a total of 20U(4U/0.1ml each)in five sites of the glabella line. Thereafter, follow-up visits will be made 4 weeks, 10weeks, 16weeks and efficacy and safety assessments will be conducted for total 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Main inclusion criteria

  1. Patients attaining ≥grade 2(moderate) in the investigator's rating of the severity of glabella line at maximum frown
* Other inclusion criteria

  1. Men and women aged between 20 and 65
  2. Patients who him/herself or him/her legal representatives voluntarily signed the informed consent
  3. Patients who can comply with the study procedures and visit schedule

Exclusion Criteria:

1. Patients with general neuromuscular synaptic disorder(e.g. Myasthenia gravis, Lambert-Eaton syndrome, Amyotrophic lateral sclerosis)
2. Patients who have bleeding tendency or taking anti-coagulant
3. Patients suffering from acute diseases
4. Patients who have been injected with botulinum toxin within past 3 months before the injection
5. Patients with allergy or hypersensitivity to the investigational products or their components
6. Patients who are pregnant or lactating or found pregnancy through the urine or serum test or disagreed to avoid pregnancy during 16 weeks study period

   * All childbearing female subjects, excepting who had amenorrhea over 12 months or sterilization operation(bilateral tubal ligation, bilateral oophorrectomy or hysterectomy), shouldn't be enrolled the study until they tested negative on pregnancy test(urine or serum). The contraceptions which are medically allowable are spermicides, oral contraceptives, barrier method, intrauterine contrace, complete sexual abstinence
7. Patients who have been given any of the following drugs within previous 4 weeks at screening

   * ① Muscle relaxants: Tubocurarine Chloride, Dantrolene Sodium, baclofen etc.
   * ② Spectinomycin HCl
   * ③ Aminoglycoside antibiotics: gentamicin sulfate, neomycin sulfate etc.
   * ④ Polypeptide antibiotics: Polymyxin B Sulfate etc.
   * ⑤ Tetracycline antibiotics
   * ⑥ Lincomycin (lincosamides)
   * ⑦ Anticholinergic drugs: butylbromide bromide, Trihexyphenidyl HCl etc.
   * ⑧ Benzodiazepines and similar drugs: Diazepam, Etizolam etc.
   * ⑨ Benzamide drugs: Tiapride HCl, Sulpiride etc.
8. Patients with the history of facial nerve paralysis or the symptoms of eyelid ptosis
9. Patients with skin damage or infection at the injection site.
10. Patients who have received or have a plan to receive other procedures which may affect glabella and forehead lines within 6 months

    * These treatments include soft tissue augmentation in the range of glabella (e.g. hyaluronic acid or collagen-type implants), medium depth peels, facial lifting, dermal photorejuvenation et cetera.
11. Patients whose glabella lines cannot be satisfactorily improved with physical method since the lines are not flattened even using hands
12. Patients who are participating in other clinical trials or have participated in other clinical trials within 30days of the screening date.
13. Patients who are unable to communicate or follow the instructions
14. Patients who are not eligible for this study at the discretion of the investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Investigator's live assessment of glabella line improvement rate | 4 weeks after the injection
  Glabella line improvement rate determined by investigator's live assessment of glabella line severity at maximum frown

SECONDARY OUTCOMES:
Investigator's live assessment of glabella line improvement rate | 16 weeks after the injection
  Glabella line improvement rate determined by investigator's live assessment of glabella line severity at maximum frown
Investigator's live assessment of glabella line improvement rate | 4, 16 weeks after the injection
  Glabella line improvement rate determined by investigator's live assessment of glabella line severity at rest.
Investigator's photographic assessment of glabella line improvement rate | 4 weeks after the injection
  Glabella line improvement rate determined by investigator's photographic assessment of glabella line severity at maximum frown
Investigator's photographic assessment of glabella line improvement rate | 4 weeks after the injection
  Glabella line improvement rate determined by investigator's photographic assessment of glabella line severity at rest.
Subject's assessment of glabella line improvement rate | 4, 10, 16 weeks after the injection
  Glabella line improvement rate determined by subject's assessment of glabella line severity.
Subject's satisfaction questionnaire | 4, 10, 16 weeks after the injection
  Subject's satisfaction of glabella line improvement at 4, 10, 16 weeks after the injection.
Number of adverse events in subjects | Up to 16 weeks
  Number of adverse events occuring in all subject for the entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: Hoon Kang, M.D., Principal Investigator — Catholic University of Korea Saint Paul's Hospital; Gwang Seong Choi, M.D., Ph.D., Principal Investigator — Inha University Hospital; Woo Young Sim, M.D., Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (3):
- South Korea (3):
  - The Catholic University of Korea, St. Paul's Hospital, Seoul, Dongdaemun-gu
  - Inha University Hospital, Incheon, Jung-gu
  - Kyung Hee University Hospital at Gangdong, Seoul, Kangdong-gu